CLINICAL TRIAL: NCT03970538
Title: Percutaneous Deep Vein Arterialization for the Treatment of Late-Stage Chronic Limb-Threatening Ischemia: the PROMISE II Trial
Brief Title: PROMISE II: Percutaneous Deep Vein Arterialization for the Treatment of Late-Stage Chronic Limb-Threatening Ischemia
Acronym: PROMISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LimFlow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LF-CA-PR-3
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Critical Limb Ischemia; Critical Lower Limb Ischemia; Peripheral Artery Disease; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Arterial Occlusive Diseases; Arterial Occlusion; Arterial Disease; Peripheral Artery Occlusion; Peripheral Vascular Disease; Peripheral Ischemia; Vascular Diseases
Keywords: CLI; CLTI; Amputation; Desert Foot; PAD; Peripheral Artery Disease; Critical Limb Ischemia; Chronic Limb-Threatening Ischemia; TADV - Transcatheter Arterialization of Deep Veins; DVA - Deep Vein Arterialization
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Arterial Occlusive Diseases; Peripheral Vascular Diseases; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center pivotal study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Treated with the LimFlow System
  Interventions: Device: LimFlow System

INTERVENTIONS:
Device: LimFlow System — Creation of an AV fistula in below-the-knee vasculature for the treatment of critical limb ischemia

SUMMARY:
The LimFlow System is intended for endovascular, minimally invasive procedures in patients who have a clinical diagnosis of chronic limb-threatening ischemia and who have been determined to have no surgical or endovascular treatment option (i.e., "no option").

DETAILED DESCRIPTION:
The objective of this US pivotal trial is to investigate the safety and effectiveness of The LimFlow System for creating an AV connection in the Below The Knee (BTK) vascular system using an endovascular, minimally invasive approach to arterialize the pedal veins for the treatment of chronic limb-threatening ischemia (CLTI) in subjects ineligible for conventional endovascular or surgical limb salvage procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 and ≤ 95 years of age
2. Clinical diagnosis of chronic limb-threatening ischemia, defined as any of the following clinical assessments: previous angiogram or hemodynamic evidence of severely diminished arterial inflow of the index limb (e.g., ABI ≤ 0.39, TP / TcPO2 < 30 mm Hg) and

   1. Rutherford Classification 5, ischemic ulceration or
   2. Rutherford Classification 6, ischemic gangrene
3. Subject has been assessed by the principal investigator, reviewed by the Independent Review Committee (IRC), and determined that no conventional distal bypass surgical or endovascular therapy for limb salvage is feasible due to either a) absence of a usable pedal artery target (endovascular or surgical approach), or b) the presence of a pedal artery target with absence of a viable single-segment vein in either lower extremity or either arm that could be used for autogenous vein conduit.
4. Proximally, the Target In-flow Artery at the cross-over point must fall within the recommended vessel diameter ranges for the LimFlow stent graft by visual estimation.
5. Prior stent(s) to the infrainguinal arteries (e.g. iliac, SFA, and popliteal) are allowed.
6. Planned minor amputation (e.g. partial toe, ray or proximal foot/transmetatarsal) of target extremity within 30 days after the index procedure is allowed.
7. Subject is willing and able to sign the informed consent form.
8. Subject is enrolled in an acceptable wound care network and has an adequate support network to ensure that subject is compliant with medication regimen and follow-up study visits.
9. Prior to enrollment (7-day window), women of childbearing potential must have a negative pregnancy test.
10. Primary wound is stable (e.g. not rapidly deteriorating and/or showing signs of healing)
11. Stable glycemic control, HbA1C < 10% (<269mg/dL)
12. Subjects requiring dialysis may be included, provided they meet all the following requirements:

    * On dialysis for > 6 months
    * Autologous arteriovenous (AV) fistula or peritoneal access used for hemodialysis
    * Serum albumin > 30 g/liter
    * BMI > 20

Exclusion Criteria:

1. Subjects will be excluded from participating in this study if they meet any of the following criteria prior to initiation of the endovascular procedure: Concomitant hepatic insufficiency, thrombophlebitis in the target limb, or non-treatable coagulation disorder within the past 90 days.
2. Active immunodeficiency disorder or currently receiving immunosuppressant therapy for an immunodeficiency disorder.
3. Prior peripheral arterial bypass procedure above or below the knee which would inhibit proximal inflow to the stent graft or interventional revascularization procedure within 30 days.
4. Previous major amputation of the target limb or presence of a wound requiring a free flap or absence of adequate viable tissue.
5. Life expectancy less than 12 months.
6. Documented myocardial infarction or stroke within previous 90 days.
7. Active infection (e.g. fever, significantly elevated WBC count >20.0 x 109/L, and/or positive blood culture) at the time of the index procedure that may preclude insertion of a prosthesis or require major amputation (e.g. osteomyelitis proximal to metatarsals).
8. Known or suspected allergies or contraindications to aspirin or P2Y12 inhibitors, heparin, stainless steel, nitinol or contrast agent that cannot be adequately pre-treated.
9. Subject is currently taking anti-coagulants, which in the opinion of the investigator, interferes with the subject's ability to participate in the study (i.e., intermittent interruption of therapy for procedure may compromise subject's safety).
10. Lower extremity vascular disease that may inhibit the procedure and/or jeopardize wound healing (e.g. vasculitis, Buerger's disease, significant edema in the target limb, deep venous thrombus in the target vein, hyperpigmentation, or medial ulceration above the ankle).
11. Significant acute or chronic kidney disease with a serum creatinine of > 2.5 mg/dl in subjects not undergoing dialysis.
12. Severe heart failure (e.g. NYHA Class IV), which in the opinion of the investigator may compromise subject's ability to safely undergo a percutaneous procedure.
13. Any significant concurrent medical, psychological, or social condition, which may significantly interfere with the subject's optimal participation in the study, in the opinion of the investigator.
14. The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.
15. 15) Subject is unwilling, or unable, or unlikely for cognitive or social reasons to comply with any of the protocol or follow-up requirements.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2025-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, MD, Principal Investigator — Vanderbilt University; Mehdi Shishehbor, Principal Investigator — University Hospital Cleveland
Locations (21):
- United States (20):
  - University of California San Francisco, San Francisco, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Yale University, New Haven, Connecticut
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Unitypoint Health, Des Moines, Iowa
  - Ochsner Health System, Kenner, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Saint Luke's Hospital, Lee's Summit, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Atrium Health, Charlotte, North Carolina
  - Coastal Carolina Surgical Associates, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Prisma Health -- Midlands, Columbia, South Carolina
  - Prisma Health -- Upstate, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Heart, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
- Ponce Medical School, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shishehbor MH, Powell RJ, Montero-Baker MF, Dua A, Martinez-Trabal JL, Bunte MC, Lee AC, Mugglin AS, Mills JL, Farber A, Clair DG; PROMISE II Investigators. Transcatheter Arterialization of Deep Veins in Chronic Limb-Threatening Ischemia. N Engl J Med. 2023 Mar 30;388(13):1171-1180. doi: 10.1056/NEJMoa2212754. PMID 36988592

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Treated with the LimFlow System
  LimFlow System: Creation of an AV fistula in below-the-knee vasculature for the treatment of critical limb ischemia
Period: Overall Study
Arm/Group | Treatment
Started | 105
Completed | 105
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 76
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 64
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Number; unit: participants]
  United States | 105
Baseline Rutherford Class 5 [Count of Participants; unit: Participants] — ISCHEMIC ULCERATION (Rutherford class 5)
  Participants | 68
Baseline Rutherford Class 6 [Count of Participants; unit: Participants] — ISCHEMIC GANGRENE (Rutherford class 6)
  Participants | 37

OUTCOME MEASURES:

1. Primary Outcome: Amputation Free Survival (AFS)
Description: freedom from major amputation and death at 6 months, compared to a historical performance goal.
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
Percentage of participants | 66

2. Secondary Outcome: Primary Patency
Description: Absence of occlusion of the endovascular intervention that is maintained without the need for additional or secondary surgical or endovascular procedures.
Time Frame: 30 days post procedure
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
percentage of participants | 68

3. Secondary Outcome: Primary Assisted Patency
Description: Absence of occlusion of the endovascular intervention maintained with the use of additional or secondary surgical or endovascular procedures, as long as occlusion of the primary treated site has not occurred.
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
Percentage of participants | 45

4. Secondary Outcome: Secondary Patency
Description: Absence of occlusion of the endovascular intervention that is maintained with the use of additional or secondary surgical endovascular procedures after occlusion occurs.
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Groups:
- Procedure Time: treated with the limflow system
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 95

5. Secondary Outcome: Limb Salvage
Description: The percentage of subjects with freedom from above-ankle amputation of the index limb.
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 94

6. Secondary Outcome: Change in Rutherford Classification
Description: A decrease in Rutherford class number (i.e.: from Rutherford class 5 to 4) is clinical improvement
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 18

7. Secondary Outcome: Technical Success
Description: The successful creation of an arteriovenous fistula in the desired limb location with immediate morphological success.
Time Frame: Immediately post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
Participants | 104

8. Secondary Outcome: Procedure Success
Description: Combination of Technical Success, and absence of all-cause death, above-ankle amputation or clinically driven major re-intervention of the stent graft.
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
Percentage of participants | 77

9. Secondary Outcome: Target Wound Healing
Description: Complete healing of the patient's target wound
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 4

10. Secondary Outcome: All Wound Healing
Description: Complete healing of the patient's wounds.
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 4

11. Secondary Outcome: Freedom From Contrast-Induced Nephropathy
Description: Subjects without acute (within 72 hours after intravenous contrast administration) impairment of renal function, measured as an absolute ≥0.5 mg/dL (44 µmol/L) increase compared to baseline SCr value that results in a value above the upper limit of the normal range.
Time Frame: Within the first 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
Participants | 103

12. Secondary Outcome: Procedure Time
Description: Time from the first puncture (venous or arterial) to when the last catheter is removed
Time Frame: Immediately post-procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
minutes | 217 (87.77)

13. Secondary Outcome: Radiation Exposure
Description: Patient radiation exposure (measured in milligray)
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: Milligray
Arm/Group | Treatment
Number analyzed (Participants) | 105
Milligray | 263 (265)

14. Secondary Outcome: Contrast Volume
Description: Total volume of contrast media (measured in milliliters)
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Treatment
Number analyzed (Participants) | 104
milliliter | 138 (80)

15. Secondary Outcome: All Wound Area Reduction
Description: Defined as reduction in area of the patient's wounds
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 11

16. Secondary Outcome: Primary Patency
Description: as for outcome 2
Time Frame: 6 months post procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 105
Percentage of participants | 26

17. Secondary Outcome: Secondary Patency
Description: as for outcome 4
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 64

18. Secondary Outcome: Limb Salvage
Description: The percentage of subjects with freedom from above-ankle amputation of the index limb.
Time Frame: 3 months days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 85

19. Secondary Outcome: Limb Salvage
Description: The percentage of subjects with freedom from above-ankle amputation of the index limb.
Time Frame: 6 months days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 76

20. Secondary Outcome: Change in Rutherford Classification
Description: A change of one Rutherford class or greater.
Time Frame: 3 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 32

21. Secondary Outcome: Change in Rutherford Classification
Description: A change of one Rutherford class or greater.
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 42

22. Secondary Outcome: Target Wound Healing
Description: Complete healing of the patient's target wound
Time Frame: 3 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 8

23. Secondary Outcome: Target Wound Healing
Description: Complete healing of the patient's target wound
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 25

24. Secondary Outcome: Target Wound Healing
Description: Complete healing of the patient's target wound
Time Frame: 9 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 37

25. Secondary Outcome: Target Wound Healing
Description: Complete healing of the patient's target wound
Time Frame: 12 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 45

26. Secondary Outcome: All Wound Area Reduction
Description: Defined as reduction in area of the patient's wounds
Time Frame: 3 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 30

27. Secondary Outcome: All Wound Area Reduction
Description: Defined as reduction in area of the patient's wounds
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 41

28. Secondary Outcome: All Wound Area Reduction
Description: Defined as reduction in area of the patient's wounds
Time Frame: 9 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 33

29. Secondary Outcome: All Wound Area Reduction
Description: Defined as reduction in area of the patient's wounds
Time Frame: 12 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 27

30. Secondary Outcome: All Wound Healing
Description: Complete healing of the patient's wounds.
Time Frame: 3 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 6

31. Secondary Outcome: All Wound Healing
Description: Complete healing of the patient's wounds.
Time Frame: 6 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 28

32. Secondary Outcome: All Wound Healing
Description: Complete healing of the patient's wounds.
Time Frame: 9 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 41

33. Secondary Outcome: All Wound Healing
Description: Complete healing of the patient's wounds.
Time Frame: 12 months post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Procedure Time
Number analyzed (Participants) | 105
Percentage of participants | 42

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 12/105
Serious Adverse Events (participants affected / at risk) | 68/105
Other Adverse Events (participants affected / at risk) | 98/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=105)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 5 (5)
Incision site impaired healing (General disorders) | 6 (6)
Gangrene (Infections and infestations) | 10 (10)
Osteomyelitis (Infections and infestations) | 7 (7)
Sepsis (Infections and infestations) | 6 (6)
Wound Infection (Infections and infestations) | 6 (6)
Wound Complication (Injury, poisoning and procedural complications) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Debridement (Skin and subcutaneous tissue disorders) | 5 (5)
Peripheral ischemia (Vascular disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=105)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Debridement (Surgical and medical procedures) | 6 (6)
Peripheral Ischemia (Vascular disorders) | 6 (6)
Impaired healing (General disorders) | 7 (7)
Incision site impaired healing (General disorders) | 6 (8)
Sepsis (Infections and infestations) | 8 (8)
Vascular stent occlusion (General disorders) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9)
Toe amputation (Surgical and medical procedures) | 9 (9)
Osteomyelitis (Infections and infestations) | 11 (11)
Wound infection (Infections and infestations) | 11 (11)
Foot amputation (Surgical and medical procedures) | 11 (11)
Wound complication (Injury, poisoning and procedural complications) | 11 (12)
Gangrene (Infections and infestations) | 12 (15)
Vascular stent occlusion (Vascular disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03970538/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT03970538/SAP_002.pdf